CLINICAL TRIAL: NCT00973960
Title: A Pilot Trial of the EndoBarrier™ Flow Restrictor for Glycemic Improvement in Type 2 Diabetics
Status: Completed | Type: Observational
Sponsor: Morphic Medical Inc. (Industry)
Responsible Party: Ken Malomo, Director of Clinical Affairs, Gi Dynamics, Inc
Other Study IDs: 09-2
Record Dates: First submitted 2009-09-06; First posted 2009-09-09 (Estimated); Last update posted 2011-08-08 (Estimated); Status verified 2011-08

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The main objective of the study is to demonstrate the safety and efficacy of the EndoBarrier Flow Restrictor in the glycemic control of diabetes in subjects with Type 2 diabetes.

The primary efficacy endpoint is an assessment of glycemic control at week 24 or last assessment measured via HbA1c.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years and < 55 years - Male or Female
* BMI > 30 BMI <60
* Subjects with an HbA1c > 7.5 and ≤ 10.0%
* Subjects with Type 2 diabetes who have been treated for ≤10 years
* Subjects on Metformin and/or Sulfonylurea
* History of failure with nonsurgical weight loss methods
* Subjects willing to comply with trial requirements
* Subjects who have signed an informed consent form
* Women who are post-menopausal, surgically sterile or on oral contraceptives and who do not plan on becoming pregnant during the course of the trial.

Exclusion Criteria:

* Treatment represents an unreasonable risk to the subject
* Subjects on oral diabetic medications other than Metformin or Sulfonylurea
* Subjects on insulin
* Subjects diagnosed with Type 1 Diabetes Mellitus or having a history of ketoacidosis
* Subjects with a past medical history of hypoglycemia
* Subjects with abnormal gastric emptying at baseline, defined as < 90% stomach emptied at 4 hours
* Subjects with a weight loss of > 4.5 Kg (10 lbs) within the 12 Weeks of screening
* Subjects taking corticosteroids or drugs known to affect GI motility (i.e. Reglan)
* Pregnant or have intention of becoming pregnant for the duration of the trial
* Unresolved alcohol or drug addiction
* Subjects receiving weight loss medications (prescription, over-the-counter, or herbal dietary medications)
* Previous gastrointestinal surgery that could affect the ability to place the EndoBarrier Flow Restrictor or the function of the implant.
* Subjects with active and uncontrolled GERD
* Subjects with symptomatic kidney stones prior to implant
* Subjects with iron deficiency and/or iron deficiency anemia
* History of Inflammatory bowel disease or condition of the gastrointestinal tract, such as ulcers or Crohn's disease
* Subjects with symptomatic gallstones prior to implant
* Symptomatic coronary artery disease or pulmonary dysfunction
* Known infection (Subjects who have a known infection at time of screening can be enrolled if the infection is treated prior to their procedure; if they still have an infection on day of procedure they must be withdrawn)
* History of congenital or acquired anomalies of the gastrointestinal tract such as atresias or stenoses
* Pancreatitis or other serious organic conditions
* Subjects requiring prescription anticoagulation therapy
* Subjects unable to discontinue NSAIDs (non-steroidal anti-inflammatory drugs) during the implant period
* Subject or Family history of a known diagnosis or pre-existing symptoms of systemic lupus erythematosus, scleroderma or other autoimmune connective tissue disorder
* Participating in another ongoing investigational clinical trial
* Mentally retarded or emotionally unstable, or exhibits psychological characteristics requiring medication that affects appetite (i.e. tricyclic antidepressants and atypical antipsychotic medications) which, in the opinion of the Investigator, makes the subject a poor candidate for device placement or clinical trial.
* Subjects with active H. pylori (Note: Subjects may be enrolled if they had a prior history of H. Pylori and were successfully treated or are diagnosed during baseline tests and undergo successful treatment before their procedure)
* Subjects with or a history of coagulopathy, upper gastro-intestinal bleeding conditions such as esophageal or gastric varices, congenital or acquired intestinal telangiectasia

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Subjects with Type 2 Diabetes
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-06 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy endpoint is an assessment of glycemic control at week 24 or last assessment measured via HbA1c. | 24 weeks

SECONDARY OUTCOMES:
The safety endpoint will be the incidence and severity of anticipated and unanticipated adverse events (device and non-device related). | 24 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Alex Escalona, MD, Principal Investigator — Hospital Universidad Catolica
Locations (1):
- Hospital Universidad Catolica, Santiago, Chile